CLINICAL TRIAL: NCT00642083
Title: Stenting of Haemodialysis Acces Re-stenosis Trial (SHARE Trial)
Brief Title: Stenting of Haemodialysis Acces Trial
Acronym: SHARE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow inclusion
Sponsor: Rijnstate Hospital (Other)
Collaborators: W.L.Gore & Associates (Industry)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: LTC-499-301107
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Outflow Stenosis
Keywords: outflow stenosis; stentgraft

ARMS (1):
- 1 (Experimental): viabahn stent-graft
  Interventions: Device: Viabahn stent-graft

INTERVENTIONS:
Device: Viabahn stent-graft — The viabahn stent-graft is a combined ePTFE-Nitinol self-expanding stent-graft preloaded on a catheter-based delivery system. It was originally designed for improving blood flow in patients with symptomatic peripheral arterial disease in superficial femoral artery lesions with reference vessel diameters ranging from 4.8 to 7.5 mm. This device is also increasingly used for the exclusion of popliteal aneurysms. Its flexibility might make the device ideal for the treatment of recurrent outflow stenosis in AV loop-fistula.

SUMMARY:
The purpose of this study is to demonstrate the efficacy of a PTFE covered stent-graft in the prevention of outflow re-stenosis in loop fistula in a prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age
* Patients have a life expectancy of at least 2 years
* Signed informed consent
* Recurrent stenosis at the venous anastomosis or in the draining vein of a loop arterio venous fistula, within 2 cm from the anastomosis.

Exclusion Criteria:

* Patient unsuitable for administration of contrast agent
* Pregnancy
* Dementia or altered mental status that would prohibit giving conscious informed consent
* Need for adjunctive major surgical or vascular procedures within one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands